CLINICAL TRIAL: NCT06894251
Title: Effect of LIMICOL®-NG on Plasma LDL-cholesterol Concentration in Subjects with Moderate Hypercholesterolemia
Acronym: LIPIGUARD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur de Lille (Other)
Responsible Party: Principal Investigator, Coralie BERTHIER, Principal Investigator, Institut Pasteur de Lille
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2024-A01916-41
Record Dates: First submitted 2025-03-11; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Healthy Volunteer
Keywords: Prevention; Food supplement; Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Intervention Model Description: Group receiving the food supplement
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Food supplement group (Experimental): Two tablets of Limicol®-NG per day (1 during or after breakfast and 1 during or after dinner) Food supplements are consumed during 3 months by healthy volunteers
  Interventions: Dietary Supplement: LIMICOL® NG

INTERVENTIONS:
Dietary Supplement: LIMICOL® NG — All subjects will consume 2 tablets per day during the entire intervention period, i.e. 12 weeks between V0 and V2, distributed as follows: 1 tablet in the morning at the end of or after breakfast (no taking on an empty stomach) and 1 tablet in the evening during dinner. If a dose is missed, 2 tablets can be taken at the next dose.

SUMMARY:
The goal of this clinical trial is to observe a decrease in plasma LDL cholesterol concentration of 10% (or 0.20g/L) in subjects with untreated moderate hypercholesterolemia after 3 months of consumption of the Limicol®-NG food supplement, compared with a historical placebo group

DETAILED DESCRIPTION:
The objective is to evaluate the effect of the Limicol®-NG food supplement during the 3 months of taking it (after 1 and 3 months of consumption versus T0) and comparison versus placebo history of the evolution over time (from 0 to 3 months) of the following parameters:

* Weight,
* BMI,
* Waist circumference,
* Systolic and diastolic blood pressures,
* Resting heart rate.
* Fasting blood sugar
* LDL cholesterol
* Non-HDL cholesterol (NHC)
* Total cholesterol (TC)
* HDL cholesterol
* Triglycerides (TG)
* LDL/HDL and TC/HDL ratios,
* Safety parameters measured from blood samples at VS and V2: ASAT, ALAT, Gamma-GT, Creatine Kinase, Lactate DeHydrogenase, Bilirubin, Creatinine, and Urea.

ELIGIBILITY:
Inclusion Criteria:

* For women

  * If pre-menopausal: effective non-estrogenic contraception established for at least 2 cycles, to be maintained during the study,
  * If menopausal: without estrogenic Hormone Replacement Therapy (HRT)
* LDL cholesterol >1.3 g/L (according to Friedewald calculation);
* Having stable eating habits, a level of physical activity and a weight for at least 3 months before the start of the study;
* Agreeing to maintain their lifestyle habits throughout the duration of the study;
* Agreeing to follow the constraints generated by the study;
* Having signed the informed consent form;
* Social security insured.

Exclusion Criteria:

* Subjects receiving hypolipidemic or anti-dyslipidemic treatment (statin, ezetimibe, cholestyramine, fibrate, etc.)
* Subjects presenting triglyceridemia > 4g/L (Friedewald)
* Subject requiring immediate treatment with statin
* Subject requiring immediate dietary intervention or having fluctuating eating behavior
* Diabetic subjects treated or not with medication
* Subjects with unstable treatment (for less than three months), or requiring the implementation of treatment during the study which, according to the investigator, could interfere with the evaluation of the study criteria (efficacy: LDL, TG, HDL, blood sugar, blood pressure, weight; safety: markers of liver, muscle or kidney function)
* Subjects who have consumed in the last 3 months food supplements or functional foods that could impact cholesterol or TG levels (phytosterol, phytostanol, red yeast rice, policosanols, beta-glucans at a dose greater than 3 g/day, probiotics)
* Subjects suffering from a severe chronic condition deemed incompatible with the study by the investigator (serious digestive pathologies, renal failure, coronary pathology, immunodeficiency, heart failure, rhythm disorders, progressive tumor pathology, blood disease)
* Subject suffering from a severe eating disorder (anorexia, bulimia, binge eating disorder)
* Pregnant woman or planning to become pregnant during the study period or breastfeeding
* Whose state of health or concomitant treatments are judged by the principal investigator or a qualified co-investigator to be incompatible with the proper conduct of the clinical study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Evolution over time (from 0 to 3 months) of the plasma concentration of LDL cholesterol | To baseline at 3 months
  Historical placebo comparison of the evolution over time (from 0 to 3 months) of plasma LDL cholesterol concentration measured according to the Friedwald method (in g/L and %).

SECONDARY OUTCOMES:
Weight | 0 month (baseline), 1 month, 3 months
  Anthropometric parameters: weight (unit: kg)
Body Mass Index | 0 month (baseline), 1 month, 3 months
  Anthropometric parameters: determined Body Mass Index (unit: kg/m²)
Waist circumference | 0 month (baseline), 1 month, 3 months
  Waist circumference (unit: cm)
Blood pressure | 0 month (baseline), 1 month, 3 months
  Hemodynamic parameters: Systolic blood pressure (unit: mm Hg) and Diastolic blood pressure (unit: mm Hg)
Heart rate | 0 month (baseline), 1 month, 3 months
  Hemodynamic parameters: Heart rate (unit: Pul/min)
Fasting glycemia | 0 month (baseline), 1 month, 3 months
  Carbohydrate metabolism: Fasting glycemia (unit: g/l)
Lipid metabolism | 0 month (baseline), 1 month, 3 months
  Total cholesterol, HDL, LDL, non-HDL, Triglycerides, LDL/HDL ratio and TC/HDL ratio (unit: g/l)
Hepatic metabolism | 0 month (baseline), 1 month, 3 months
  Creatinine, bilirubin (unit: mg/dl)
Transaminases | 0 month (baseline), 1 month, 3 months
  Hepatic metabolism: ASAT/ALAT, GGT (unit: UI/l)
Renal metabolism (Urea) | 0 month (baseline), 1 month, 3 months
  Renal metabolism: Urea (unit: mg/dl)
Renal metabolism (Creatinine Phophoskinase) | 0 month (baseline), 1 month, 3 months
  Renal metabolism: CPK (unit : UI/l)
Renal metabolism (Lactate Deshydrogenase) | 0 month (baseline), 1 month, 3 months
  Renal metabolism: LDH (unit : UI/l)

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Batteux, MD, Principal Investigator — Institut Pasteur de Lille
Locations (1):
- NutrInvest - Institut Pasteur de Lille, Lille, Nord, France